CLINICAL TRIAL: NCT05187741
Title: Effect of an Mobile Health Intervention on Adherence to Antiretroviral Treatment in Adult Patients Living With HIV Compared to Standard Care
Brief Title: Effect of a Mobile Health Intervention on Treatment Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, Luis Eduardo del Moral Trinidad, Public Health Master Student, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 138/21
Record Dates: First submitted 2021-12-13; First posted 2022-01-12 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: HIV I Infection
Keywords: electronic health; adherence

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily message group (Experimental): This group would be receiving text messages intended to improve treatment adherence and text reminders for appointments to improve care retention.
  Interventions: Device: mobile health (mHealth)
- Control group (No Intervention): This group would be just observed through the same period as the intervention group but the participants will only receive the standard care provide by the clinic.

INTERVENTIONS:
Device: mobile health (mHealth) — A message will be sent on Monday and Friday at 9:00 am for 3 months, the first day they will receive a message focused on adherence and the second day a message focused on motivation. Subsequently, a message will be sent on Mondays for 3 more months.
  Reminders for appointments with your treating physician will be sent during the entire intervention period (6 months).
  Arms: Daily message group

SUMMARY:
This is a randomized clinical trial across the whole of the patients who attend the HIV Unit of the Hospital Civil Viejo, a sample calculated in 43 patients for each group (intervention and control). Patients who have HIV infection and are starting antiretroviral treatment (ART), who are between 18 and 50 years old and have a mobile device, will be included in the study. The messages will consist of medical appointment reminders and adherence and motivational messages for a period of six months.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with HIV infection

  . starting with antiretroviral therapy and haven't taken ART before
* Patients with the status of "lost to follow up" who return to re-initiate ART

Exclusion Criteria:

* Patients who are participating in other study
* patients above 18 years old
* Patients who does not have signal phone at their residency
* Those who refuses to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
antiretroviral treatment adherence | 6 months
  The practice of patients where they take their medications as prescribed. To proceed with the calculation, the following formula should be applied: [(number of units dispensed - number of units remaining) / (prescribed number of units per day x number of days between the two visits)] x 100.

SECONDARY OUTCOMES:
care retention | 6 months
  Person living with HIV who enters and remains in comprehensive HIV care by health services, according to their needs. It is recorded at 6 months and 12 months of follow-up, with the patient's compliance with their medical appointments.
HIV viral loal | 6 months
  Amount of genetic material (RNA) of the virus in blood in the most recent determination.Measure by Reverse transcriptase polymerase chain reaction test reported as copies/ml
TCD4+ count in blood | 6 months
  Number of CD4 + T lymphocytes in the blood. Measure by flow cytometry and reported as cells/mm3

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No